CLINICAL TRIAL: NCT01076933
Title: Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) on Borderline Personality Disorder (BPD)
Brief Title: Transcranial Magnetic Stimulation for Borderline Personality Disorder
Acronym: SiMaT-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08 153 02; AOL 2008
Record Dates: First submitted 2010-01-06; First posted 2010-02-26 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Transcranial Magnetic Stimulation; Neuropsychological Test; Randomised Control Trial
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS (Experimental): rTMS sessions
  Interventions: Procedure: repetitive Transcranial Stimulation Magnetic (rTMS)
- control (Sham Comparator): sham rTMS (control)
  Interventions: Procedure: sham rTMS

INTERVENTIONS:
Procedure: repetitive Transcranial Stimulation Magnetic (rTMS) — The motor threshold was determined in each subject once, before treatment. This was defined as the lowest stimulation intensity capable of inducing a visible movement at least five times out of 10 stimulations. The position of the right dorsolateral prefrontal cortex was defined as 5 cm anterior (in a parasagittal line) to the motor cortex. The stimulus intensity was 80% of the patient's motor threshold intensity. Treatments were given for 20 minutes per day over 10 working days.
  Arms: rTMS
Procedure: sham rTMS — sham rTMS
  Arms: control

SUMMARY:
Primary purpose : to assess the effect on neuropsychological tasks related to planning of 10 daily sessions of right dorsolateral prefrontal cortex with High-frequency repetitive transcranial magnetic stimulation (rTMS) on borderline personality disorder (BPD) patients.

Hypothesis : BPD patients receiving 10 sessions of rTMS will have greater improvement in the average number of move to achieve tasks of the Tower of London, than those receiving sham rTMS.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 45 years old
* Borderline Personality Disorder (Diagnostic Interview for Borderline Personality Disorder > 8)
* psychiatric follow-up
* righthander
* informed consent
* affiliated to medical insurance

Exclusion Criteria:

* bipolar disorder
* substance use disorder
* Major Depressive Disorder or Stress Post Traumatic Disorder
* history of epilepsy
* neurosurgery
* cardiac pacemaker
* lefthander
* involuntary admission
* participation in an other research
* legal guardianship
* poor mastery of french.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Tower of London | Inclusion, 15th day, 30th day and 3rd month

SECONDARY OUTCOMES:
Balloon Analog Risk Task | Inclusion, 15th day, 30th day and 3rd month
Micro-World Test | Inclusion, 15th day and 3rd month
Borderline Personality Disorder Severity Index | Pre-inclusion, 30th day and 3rd month
Symptom Check List - 90 | Inclusion, 15th day, 30th day and 3rd month
Barratt Impulsivity Scale | Inclusion and 3rd month
Global Assessment Scale | Inclusion and 3rd month

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Cailhol, MD, Principal Investigator — University Hospital Toulouse - 31059 Toulouse - France
Locations (1):
- Lionel Cailhol, Toulouse, University Hospital Toulouse, France

REFERENCES:
- [Result] Cailhol L, Roussignol B, Klein R, Bousquet B, Simonetta-Moreau M, Schmitt L, Thalamas C, Tap G, Birmes P. Borderline personality disorder and rTMS: a pilot trial. Psychiatry Res. 2014 Apr 30;216(1):155-7. doi: 10.1016/j.psychres.2014.01.030. Epub 2014 Jan 30. PMID 24503285